CLINICAL TRIAL: NCT03514602
Title: Pilot Study on Pediatric Obesity Prevention by Maternal Smoking Cessation in Pregnancy and Lactation
Brief Title: Maternal Smoking Cessation and Pediatric Obesity Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Xiaozhong Wen, Assistant Professor, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MODCR00001304
Record Dates: First submitted 2018-01-22; First posted 2018-05-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Childhood Obesity; Smoking, Cigarette; Pregnancy
MeSH Terms: conditions — Pediatric Obesity; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Multicomponent behavioral intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent behavioral intervention (Experimental): The multicomponent intervention group will receive education and counseling, monitoring and feedback, contingent financial incentives, and family support.
  Interventions: Behavioral: Multicomponent behavioral intervention
- Control (Active Comparator): The control group will receive smoking cessation education only.
  Interventions: Behavioral: Education only control

INTERVENTIONS:
Behavioral: Multicomponent behavioral intervention — Pregnant patients in the intervention group will receive multicomponent interventions consisting of education, feedback, contingent financial incentives, and peer support. At initial intervention visit, they will choose a quit date within the next 14 days and sign a no-smoking pledge and a no-smoking contract. The contract lists the intervention components, the patient's and the counselor's responsibilities, importance of keeping scheduled visits, and rules on contingent incentives. After the quit date, pregnant women will meet with counselors daily for 5 consecutive days (Monday to Friday) for abstinence monitoring in weeks 1-2. The frequency of abstinence monitoring will decrease to twice a week (Monday and Thursday) in weeks 3-8, weekly in weeks 9-12, and biweekly in weeks 13 until delivery.
  Arms: Multicomponent behavioral intervention
Behavioral: Education only control — The control group will receive one 60-minute counseling mainly based on a pregnancy-tailored self-help booklet entitled "Need Help Putting Out That Cigarette?" distributed by the American College of Obstetricians and Gynecologists.
  Arms: Control

SUMMARY:
The objective of this study is to test the effect of smoking cessation in pregnancy or in lactation on preventing rapid infant adiposity gain. Investigators propose a randomized, controlled experiment among smoking pregnant women from 1st prenatal care visit through 6 months of postpartum period. Two-phase randomization will be applied to separate the effects of smoking cessation in two different critical periods (i.e., pregnancy and lactation) on infant adiposity gain. Investigators will first randomly assign 40 smoking pregnant women into either the multicomponent intervention (N=30) or the education-only control group (N=10). The multicomponent intervention group will receive education and counseling, monitoring and feedback, contingent financial incentives, and family support, while the control group will receive education only. At the end of pregnancy, investigators will further randomize successful quitters (estimated N=20) from the multi-component intervention group into either the continuous multi-component intervention group in lactation (N=10) or the education-only control group (N=10). All women and their newborns will be followed from enrollment to 6 months postpartum. The key outcomes include maternal smoking abstinence confirmed by urine-cotinine and infant gain in weight-for-length z-score. Specific Aim 1 is to examine the effects of maternal smoking cessation intervention in pregnancy on infant gain in weight-for-length z-score from birth to 6 months. Specific Aim 2 is to examine the effect of maternal smoking abstinence intervention in lactation and infant post-weaning gain in weight-for-length z-score among the women who have successfully quit smoking in pregnancy.

DETAILED DESCRIPTION:
The objective of this study is to test the effect of smoking cessation in pregnancy or in lactation on preventing rapid infant adiposity gain. Investigators propose a randomized, controlled experiment among smoking pregnant women from 1st prenatal care visit through 6 months of postpartum period. Two-phase randomization will be applied to separate the effects of smoking cessation in two different critical periods (i.e., pregnancy and lactation) on infant adiposity gain. Investigators will first randomly assign 40 smoking pregnant women into either the multicomponent intervention (N=30) or the education-only control group (N=10). The multicomponent intervention group will receive education and counseling, monitoring and feedback, contingent financial incentives, and family support, while the control group will receive education only. At the end of pregnancy, investigators will further randomize successful quitters (estimated N=20) from the multi-component intervention group into either the continuous multi-component intervention group in lactation (N=10) or the education-only control group (N=10). All women and their newborns will be followed from enrollment to 6 months postpartum.The key outcomes include maternal smoking abstinence confirmed by urine-cotinine and infant gain in weight-for-length z-score. Specific Aim 1 is to examine the effects of maternal smoking cessation intervention in pregnancy on infant gain in weight-for-length z-score from birth to 6 months. Specific Aim 2 is to examine the effect of maternal smoking abstinence intervention in lactation and infant post-weaning gain in weight-for-length z-score among the women who have successfully quit smoking in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and speak English.
2. Are 18-39 years old
3. Are less than 20 weeks of gestation
4. Have a singleton pregnancy
5. Currently smoking one or more cigarettes per day, based on self-report.
6. Currently smoking biochemically verified by a level of 1 or higher in urine cotinine test (i.e., >100ng/mL cotinine concentration).
7. Willing to try to quit or reduce smoking by behavioral intervention
8. Willing to monitor smoking status by breath carbon monoxide and saliva cotinine.
9. Willing to provide breath, saliva, and urine samples to test smoking status
10. With low household income (meeting federal income eligibility guidelines for the Special Supplemental Nutrition Program for Women, Infants, and Children) and/or low education level (≤12 years). These disadvantaged pregnant women are very likely not to quit spontaneously, and thus need extra intervention most.
11. Currently living in Erie County or Niagara County; don't plan to move out of these two counties during the current pregnancy.

Exclusion Criteria:

1. Previous history of major chronic disease or blood clotting disorders such as cancer, thyroid disorders, heart disease, kidney disease
2. Depression or have been diagnosed with depression or post-partum depression at any time
3. In treatment for Axis 1 disorders that prevent them following smoking cessation interventions

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported Smoking abstinence verified by urine cotinine test | At end of pregnancy (35 weeks of pregnancy; an average of 10 weeks after intervention)
  Self-reported Smoking abstinence verified by urine cotinine test

SECONDARY OUTCOMES:
Infant gain in weight-for-length z-score | from birth to 12 months
  Infant gain in weight-for-length z-score

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Wen, MD, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Division of Behavioral Medicine Department of Pediatrics Jacobs School of Medicine and Biomedical Sciences State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No